CLINICAL TRIAL: NCT05580276
Title: Investigation of Temporamandibular Joint Functions and Parafunctional Habits in Adolescents With Headache
Brief Title: Temporamandibular Joint Functions and Parafunctional Habits
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Nurhayat KORKMAZ, Research assistant, Karadeniz Technical University
Other Study IDs: KTU-FTR-02
Record Dates: First submitted 2022-09-28; First posted 2022-10-14 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Headache; Temporomandibular Disorder
Keywords: adolescent headache; temporomandibular dysfunction
MeSH Terms: conditions — Headache; Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Adolescent with headache, 10-18 ages
- Control group: Adolescent without headache

SUMMARY:
Headache is the most common type of pain in children and adolescents with effects on health-related quality of life (HrQoL), school attendance, and social functioning. The International Headache Society recognizes that secondary headaches can be attributed to temporamandibular joint (TMJ) problems. The primary aim of the study is to evaluate temporamandibular joint functions and parafunctional habits in adolescents with headache. The second aim is to examine the relationship between temporamandibular joint functions and parafunctional habits and headache.

DETAILED DESCRIPTION:
24 individuals under the age of 18 diagnosed with headache and 24 healthy controls will be included in the study. Age, height, weight characteristics and parafunctional habits of individuals will be recorded. The severity of headache and its effect on daily life, temporamandibular joint pain severity will be evaluated. Temporamandibular joint dysfunction severity will be determined and mouth openings will be measured.

Participants who meet the inclusion criteria will be included in the study group. Healthy volunteers without headache complaints will also be included in the study as a control group.In this study, which is planned to include those who meet the inclusion criteria and agree to participate in the study, written informed consent form will be obtained from all individuals and from their parents for those under the age of 18. The study will be carried out in accordance with the ethical principles of the Declaration of Helsinki. The study will be done through a questionnaire form and with anthropetric measurements. No invasive procedure will be applied. A p value of ≤0.05 will be considered significant in all statistics.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with headache according to the ICDH-II (International Classification of Headache Disorders 2nd edition) criteria published by IHS (International Headache Society) in 2004
* Having a headache complaint in the last 3 months
* Having a HIT-6 score of 50 or higher

Exclusion Criteria:

* Being on any analgesic, anti-sedative, myorelaxant medication
* Those with mental and psychiatric problems

Ages: 10 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Adolescents 10-18 years old with headache and without headache
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Headache Impact Test (HIT-6) | 1 day (one assessment)
Temporomandibular dysfunction | 1 day (one assessment)
  Fonseca Anamnestic Index. No dysfunction, mild, moderate, severe

SECONDARY OUTCOMES:
Wong Baker Pain Scale | 1 day (one assessment)
  Severity of Headache
Mouth opening measurement | 1 day (one assessment)
  Maximum painless mouth opening width and lateral deviations from the distance between the two anterior incisors in the lower and upper palate
Pressure pain threshold | 1 day (one assessment)
  Pressure pain thresholds of temporomandibular joint, masseter, temporalis, SCM and upper trapezius muscles
Parafunctional habits questionnaire | 1 day (one assessment)
  Teeth clenching, teeth grinding, lip biting, excessive gum chewing, pencil biting, nail biting, hands on chin, chewing on one side only, sleeping on one side only

CONTACTS AND LOCATIONS:
Overall Officials: Elif Acar Arslan, Assoc. Prof, Study Director — Karadeniz Technical University
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No